CLINICAL TRIAL: NCT01998464
Title: Evaluation of the Utility of OCT Angiography in Assessing Vascular Perfusion in Retinal Vasculitis
Brief Title: Optical Coherence Tomography (OCT) in Retinal Vasculitis
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Phoebe Lin, MD, PhD, Assistant Professor of Ophthalmology, Oregon Health and Science University
Other Study IDs: OHSU IRB#00010137
Record Dates: First submitted 2013-11-18; First posted 2013-11-29 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Retinal Vasculitis
Keywords: Retinal Vasculitis; Optical coherence tomography; OCT; Imaging
MeSH Terms: conditions — Retinal Vasculitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Retinal Vasculitis Group: Up to 35 patients diagnosed with retinal vasculitis will be considered and evaluated for enrollment in this study.

SUMMARY:
Retinal vasculitis is a sight-threatening inflammation that involves the blood vessels of the retina, the tissue that lines the inside of the eye. This inflammation may occur on its own or as a result of an infectious, cancerous, or inflammatory disorder.

Optical coherence tomography (OCT) is an imaging technology that can perform non-contact cross-sectional imaging of retinal and choroidal tissue structure in real time. It is similar to ultrasound imaging, except that OCT measures the intensity of reflected light rather than sound waves.

The purpose of this study is to see if non-invasive OCT technology can diagnose retinal vasculitis as well as the more invasive fluorescein angiography, which requires an injection of dye into the vein of an arm of a patient. The study will also compare the mapping of blood vessels (angiography) and loss of blood flow (ischemia) by fluorescein angiography and OCT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of retinal vasculitis

Exclusion Criteria:

* Inability to give informed consent.
* Inability to complete the qualifying study tests within a 30 day period from date of enrollment
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A prior history of reaction to fluorescein or other dyes.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g. unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, subject can become eligible.
* Systemic anti-vascular endothelial growth factor (VEGF) or pro-VEGF treatment within 4 months prior to treatment.
* Women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months due to unknown safety of fluorescein angiography.
* Prior panretinal photocoagulation (PRP) or focal laser that would alter the macular perfusion and retinovascular features.
* Inability to maintain stable fixation for OCT imaging.
* Other ocular condition is present such that, in the opinion of the investigator, may alter the retinal perfusion.
* An ocular condition is present that, in the opinion of the investigator, might affect or alter visual acuity during the course of the study (i.e. cataract)
* Substantial cataract that, in the opinion of the investigator, is likely to decrease visual acuity by 3 lines or more (i.e. cataract would be reducing acuity to 20/40 or worse if the eye was otherwise normal).
* Media opacity or otherwise that would prevent either fixation or ability to obtain adequate images as determined by the examiner.
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc) within prior 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will measure blood vessel pattern/flow changes in up to 35 patients with retinal vasculitis.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Blood flow patterns in retinal vasculitis | 24 months
  To determine if identifying early changes in blood vessel patterns will aid in early diagnosis and treatment of retinal vasculitis. Total retinal blood flow will be measured in uL/min.

SECONDARY OUTCOMES:
Ischemia in retinal vasculitis | 24 months
  To determine if identifying lost or reduced blood flow will aid in early diagnosis and treatment of retinal vasculitis. Non-perfusion area will be measured in mm2.

CONTACTS AND LOCATIONS:
Overall Officials: Phoebe Lin, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States